CLINICAL TRIAL: NCT00416377
Title: Hodgkin's Disease Study
Brief Title: Radiation Therapy or Combination Chemotherapy in Treating Young Patients With Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-HD-9201; CDR0000454741 (Registry Identifier: PDQ (Physician Data Query)); EU-20586
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-12

CONDITIONS: Lymphoma
Keywords: stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Bleomycin; Chlorambucil; Dacarbazine; Doxorubicin; Prednisolone; Procarbazine; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: chlorambucil
Drug: dacarbazine
Drug: doxorubicin hydrochloride
Drug: prednisolone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill cancer cells. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This clinical trial is studying how well radiation therapy or combination chemotherapy work in treating young patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Maintain the present satisfactory results of patients treated on protocol UKCCSG-HD-8201 in pediatric patients with stage I-III Hodgkin's lymphoma treated with radiotherapy or combination chemotherapy comprising chlorambucil, procarbazine hydrochloride, prednisolone, vinblastine followed by doxorubicin hydrochloride, bleomycin, vincristine, and dacarbazine.
* Determine, by comparison with UKCCSG-HD-8201, if mediastinal irradiation can be safely omitted from the management of pediatric patients with Hodgkin's lymphoma and bulky mediastinal disease.
* Determine if gallium scanning of the mediastinum after chemotherapy will identify patients with residual active mediastinal disease.
* Improve disease control in patients with stage IV Hodgkin's lymphoma and slow responders by intensifying treatment to patients who fail to achieve complete remission after 4 courses of chlorambucil, vinblastine, procarbazine hydrochloride, and prednisone.

OUTLINE: This is a multicenter study. Patients are stratified according to stage of disease (I vs II-IV).

* Stage I: Patients undergo involved-field radiotherapy.
* Stage II-IV:

  * CHLVPP chemotherapy: Patients receive CHLVPP chemotherapy comprising oral chlorambucil, oral procarbazine hydrochloride, and oral prednisolone on days 1-14 and vinblastine IV on days 1-8. Treatment repeats every 28 days for 2 courses. Patients achieving complete resolution (CR) of measurable disease receive an additional 4 courses of CHLVPP. Patients with no response or progressive disease proceed to ABVD chemotherapy. Patients with shrinkage of measurable disease to < 50% original dimensions (GPR) receive 2 additional courses of CHLVPP. Patients achieving CR or GPR after completion of 2 additional courses of CHLVPP receive 4 more courses of CHLVPP. Patients achieving shrinkage of measurable disease to ≥ 50% of original dimension (PR) after 2 additional courses of CHLVPP OR patients not achieving CR after a total of 8 courses of CHLVPP proceed to ABVD chemotherapy.
  * ABVD chemotherapy: Patients receive ABVD chemotherapy comprising doxorubicin hydrochloride IV over 4 hours and bleomycin IV, vincristine IV, and dacarbazine IV on days 1 and 15. Treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
* Mediastinal mass: Patients receive chemotherapy as per stages II-IV. Patients presenting with airway or superior vena cava obstruction may also undergo radiotherapy. Patients achieving CR after completion of chemotherapy receive no further treatment. Patients achieving GPR or PR after completion of chemotherapy undergo gallium scan and CT scan of thorax with or without biopsy at the investigator's discretion.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 353 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed childhood Hodgkin's lymphoma by lymph node biopsy

  * Any stage disease
  * Patients with bilateral upper cervical disease with no evidence of supraclavicular, thoracic inlet, or Waldeyers ring involvement are treated as having stage I disease

PATIENT CHARACTERISTICS:

* Platelet count > 100,000/mm^3
* Absolute neutrophil count > 1,000/mm^3

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Barrett, Study Chair — University of Glasgow; Judith E. Kingston, MD — St. Bartholomew's Hospital; John Martin, MD — Royal Liverpool Children's Hospital, Alder Hey